CLINICAL TRIAL: NCT02564900
Title: Phase 1, Two-Part, Multicenter, Non-randomized, Open-label, Multiple Dose First-In-Human Study of DS-8201A, in Subjects With Advanced Solid Malignant Tumors
Brief Title: Study of DS-8201a in Subjects With Advanced Solid Malignant Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Daiichi Sankyo Co., Ltd. (Industry)
Collaborators: Daiichi Sankyo (Industry); AstraZeneca (Industry)
Responsible Party: Sponsor
Organization: Daiichi Sankyo (Industry)
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: DS8201-A-J101; 152978 (Registry Identifier: JAPIC CTI)
Record Dates: First submitted 2015-09-21; First posted 2015-10-01 (Estimated); Results first posted 2021-06-23 (Actual); Last update posted 2024-01-22 (Actual); Status verified 2024-01

CONDITIONS: Advanced Solid Tumors
Keywords: Advanced solid tumors; phase 1; oncology; HER2; Antibody drug conjugate (ADC)
MeSH Terms: conditions — Neoplasms | interventions — trastuzumab deruxtecan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Part 1 Dose escalation (Experimental): Part 1 is a dose escalation to identify the Maximum Tolerated dose (MTD) or the recommended phase 2 dose of DS-8201a guided by the modified continuous reassessment method using a Bayesian logistic regression model following escalation with overdose control principal.
  Interventions: Drug: DS-8201a (DP1); Drug: DS-8201a (DP)
- Part 2 Dose expansion (Experimental): Part 2 is a dose expansion to examine the safety and efficacy of DS-8201a and it is consist of multiple cohorts: in subjects with trastuzumab emtansine (T-DM1)-treated HER2 overexpressing breast cancer (Part 2a); trastuzumab-treated HER2 overexpressing gastric or gastroesophageal junction adenocarcinoma (Part 2b); HER2 low expressing breast cancer (Part 2c), HER2 expressing other solid malignant tumor (Part 2d); HER2 expressing breast cancer (Japan only; Part 2e)
  Interventions: Drug: DS-8201a (DP1); Drug: DS-8201a (DP2); Drug: DS-8201a (DP)

INTERVENTIONS:
Drug: DS-8201a (DP1) — DS-8201a to be administered via intravenous (IV) dose. DS-8201a (DP1) was used for the Dose Escalation phase and for Dose expansion Parts 2a, 2b, 2c, and 2d.
Drug: DS-8201a (DP2) — DS-8201a is to be administered via intravenous (IV) dose. DS-8201a (DP2) was used only used for Dose Expansion Part 2e.
  Arms: Part 2 Dose expansion
Drug: DS-8201a (DP) — DS-8201a (DP) is to be administered via intravenous (IV) dose.

SUMMARY:
This is an open-label, two-part, multicenter study to evaluate the safety and tolerability of DS-8201a in participants with advanced solid malignant tumors.

ELIGIBILITY:
Inclusion Criteria:

* Eastern Cooperative Oncology Group performance status( PS) of 0 or 1.
* Left Ventricular Ejection Fraction (LVEF) ≥ 50%

Part 1:

* Advanced/unresectable or metastatic breast cancer or gastric or gastroesophageal junction adenocarcinoma that is refractory to or intolerable with standard treatment, or for which no standard treatment is available.

Part 2a:

* Advanced breast cancer with HER2 overexpression that is refractory to or intolerable with standard treatment, or for which no standard treatment is available.
* Treated with ado-trastuzumab emtansine (T-DM1)

Part 2b:

* Advanced gastric or gastroesophageal junction adenocarcinoma with HER2 overexpression that is refractory to or intolerable with standard treatment, or for which no standard treatment is available.
* Treated with trastuzumab

Part 2c:

* Advanced breast cancer with HER2 low expression that is refractory to or intolerable with standard treatment, or for which no standard treatment is available.

Part 2d:

* Satisfy at least one of the following criteria

  1. Advanced/unresectable or metastatic solid malignant tumor with HER2 expression other than breast cancer and gastric or gastroesophageal junction adenocarcinoma that is refractory to or intolerable with standard treatment, or for which no standard treatment is available.
  2. Advanced/unresectable or metastatic tumor with HER2 mutation that is refractory to or intolerable with standard treatment, or for which no standard treatment is available.

Part 2e:

* Advanced breast cancer with HER2 overexpression that is refractory to or intolerable with standard treatment, or for which no standard treatment is available.
* Treated with ado-trastuzumab emtansine (T-DM1) (patients with HER2 overexpression only)

Exclusion Criteria:

* Has a medical history of symptomatic Congestive Heart Failure (CHF) (NYHA classes II-IV) or serious cardiac arrhythmia.
* Has a medical history of myocardial infarction or unstable angina.
* Has a QTc prolongation to > 450 millisecond (ms) in males and > 470 ms in females.
* Has a medical history of clinically significant lung diseases

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 292 (Actual)
Dates: Start 2015-09-01 (Actual); Primary Completion 2019-02-01 (Actual); Study Completion 2023-12-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Leader, Study Director — Daiichi Sankyo
Locations (14):
- United States (8):
  - Sharp Memorial Hospital, San Diego, California
  - Mayo Clinic, Jacksonville, Florida
  - University of Louisville, Louisville, Kentucky
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Washington University School of Medicine, St Louis, Missouri
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - UC Health Clinical Trials Office, Cincinnati, Ohio
  - University of Texas M. D. Anderson Cancer Center, Houston, Texas
- Japan (6):
  - Aichi Cancer Center Hospital, Aichi
  - National Cancer Center Hospital East, Chiba
  - Social Medical Corporation Hakuaikai Sagara Hospital, Kagoshima
  - Kindai University Hospital, Osaka
  - National Cancer Center Hospital, Tokyo
  - The Cancer Institute Hospital of Japanese Foundation For Cancer Research, Tokyo

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD) and applicable supporting clinical trial documents may be available upon request at https://vivli.org/. In cases where clinical trial data and supporting documents are provided pursuant to our company policies and procedures, Daiichi Sankyo will continue to protect the privacy of our clinical trial participants. Details on data sharing criteria and the procedure for requesting access can be found at this web address: https://vivli.org/ourmember/daiichi-sankyo/
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Studies for which the medicine and indication have received European Union (EU) and United States (US), and/or Japan (JP) marketing approval on or after 01 January 2014 or by the US or EU or JP Health Authorities when regulatory submissions in all regions are not planned and after the primary study results have been accepted for publication.
Access Criteria: Formal request from qualified scientific and medical researchers on IPD and clinical study documents from clinical trials supporting products submitted and licensed in the United States, the European Union and/or Japan from 01 January 2014 and beyond for the purpose of conducting legitimate research. This must be consistent with the principle of safeguarding study participants' privacy and consistent with provision of informed consent.
URL: https://vivli.org/ourmember/daiichi-sankyo/

REFERENCES:
- [Result] Tsurutani J, Iwata H, Krop I, Janne PA, Doi T, Takahashi S, Park H, Redfern C, Tamura K, Wise-Draper TM, Saito K, Sugihara M, Singh J, Jikoh T, Gallant G, Li BT. Targeting HER2 with Trastuzumab Deruxtecan: A Dose-Expansion, Phase I Study in Multiple Advanced Solid Tumors. Cancer Discov. 2020 May;10(5):688-701. doi: 10.1158/2159-8290.CD-19-1014. Epub 2020 Mar 25. PMID 32213540
- [Result] Tamura K, Tsurutani J, Takahashi S, Iwata H, Krop IE, Redfern C, Sagara Y, Doi T, Park H, Murthy RK, Redman RA, Jikoh T, Lee C, Sugihara M, Shahidi J, Yver A, Modi S. Trastuzumab deruxtecan (DS-8201a) in patients with advanced HER2-positive breast cancer previously treated with trastuzumab emtansine: a dose-expansion, phase 1 study. Lancet Oncol. 2019 Jun;20(6):816-826. doi: 10.1016/S1470-2045(19)30097-X. Epub 2019 Apr 29. PMID 31047803
- [Result] Shitara K, Iwata H, Takahashi S, Tamura K, Park H, Modi S, Tsurutani J, Kadowaki S, Yamaguchi K, Iwasa S, Saito K, Fujisaki Y, Sugihara M, Shahidi J, Doi T. Trastuzumab deruxtecan (DS-8201a) in patients with advanced HER2-positive gastric cancer: a dose-expansion, phase 1 study. Lancet Oncol. 2019 Jun;20(6):827-836. doi: 10.1016/S1470-2045(19)30088-9. Epub 2019 Apr 29. PMID 31047804
- [Result] Modi S, Saura C, Yamashita T, Park YH, Kim SB, Tamura K, Andre F, Iwata H, Ito Y, Tsurutani J, Sohn J, Denduluri N, Perrin C, Aogi K, Tokunaga E, Im SA, Lee KS, Hurvitz SA, Cortes J, Lee C, Chen S, Zhang L, Shahidi J, Yver A, Krop I; DESTINY-Breast01 Investigators. Trastuzumab Deruxtecan in Previously Treated HER2-Positive Breast Cancer. N Engl J Med. 2020 Feb 13;382(7):610-621. doi: 10.1056/NEJMoa1914510. Epub 2019 Dec 11. PMID 31825192
- [Result] Doi T, Shitara K, Naito Y, Shimomura A, Fujiwara Y, Yonemori K, Shimizu C, Shimoi T, Kuboki Y, Matsubara N, Kitano A, Jikoh T, Lee C, Fujisaki Y, Ogitani Y, Yver A, Tamura K. Safety, pharmacokinetics, and antitumour activity of trastuzumab deruxtecan (DS-8201), a HER2-targeting antibody-drug conjugate, in patients with advanced breast and gastric or gastro-oesophageal tumours: a phase 1 dose-escalation study. Lancet Oncol. 2017 Nov;18(11):1512-1522. doi: 10.1016/S1470-2045(17)30604-6. Epub 2017 Oct 13. PMID 29037983
- [Derived] Takahashi S, Bando H, Kinoshita I, Modi S, Tsurutani J, Bang YJ, Sato Y, Nakatani S, Lee C, Sugihara M, Okuda Y, Iwata H. Trastuzumab deruxtecan in patients with human epidermal growth factor receptor 2-expressing salivary gland carcinoma: a pooled analysis of two phase I studies. Jpn J Clin Oncol. 2024 Apr 6;54(4):434-443. doi: 10.1093/jjco/hyad181. PMID 38231777
- [Derived] Yin O, Iwata H, Lin CC, Tamura K, Watanabe J, Wada R, Kastrissios H, AbuTarif M, Garimella T, Lee C, Zhang L, Shahidi J, LaCreta F. Exposure-Response Relationships in Patients With HER2-Positive Metastatic Breast Cancer and Other Solid Tumors Treated With Trastuzumab Deruxtecan. Clin Pharmacol Ther. 2021 Oct;110(4):986-996. doi: 10.1002/cpt.2291. Epub 2021 Jun 10. PMID 33999422
- [Derived] Modi S, Park H, Murthy RK, Iwata H, Tamura K, Tsurutani J, Moreno-Aspitia A, Doi T, Sagara Y, Redfern C, Krop IE, Lee C, Fujisaki Y, Sugihara M, Zhang L, Shahidi J, Takahashi S. Antitumor Activity and Safety of Trastuzumab Deruxtecan in Patients With HER2-Low-Expressing Advanced Breast Cancer: Results From a Phase Ib Study. J Clin Oncol. 2020 Jun 10;38(17):1887-1896. doi: 10.1200/JCO.19.02318. Epub 2020 Feb 14. PMID 32058843
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/32213540/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 292 participants who met all inclusion and no exclusion criteria were enrolled at 8 centers in the US and 6 centers in Japan. A total of 27 participants started the Dose Escalation phase and a total of 265 participants in the Dose Expansion phase.
Pre-assignment Details: The Dose Escalation was intended to identify the maximum tolerated dose (MTD) or recommended phase 2 dose (RP2D) of DS-8201a with at least 3 participants evaluable for assessment of dose-limiting toxicity per dose level. Since the MTD was not reached, doses of 5.4 mg/kg and 6.4 mg/kg were chosen for evaluation in the Dose Expansion phase.
Groups:
- Dose Escalation: Cohort 1, 0.8 mg/kg: Participants in Cohort 1 received an intravenous 0.8 mg/kg dose of DS-8201a (FL-DP1).
- Dose Escalation: Cohort 2, 1.6 mg/kg: Participants in Cohort 2 received an intravenous 1.6 mg/kg dose of DS-8201a (FL-DP1).
- Dose Escalation: Cohort 3, 3.2 mg/kg: Participants in Cohort 3 received an intravenous 3.2 mg/kg dose of DS-8201a (FL-DP1).
- Dose Escalation: Cohort 4, 5.4 mg/kg: Participants in Cohort 4 received an intravenous 5.4 mg/kg dose of DS-8201a (FL-DP1).
- Dose Escalation: Cohort 5, 6.4 mg/kg: Participants in Cohort 5 received an intravenous 6.4 mg/kg dose of DS-8201a (FL-DP1).
- Dose Escalation: Cohort 6, 8.0 mg/kg: Participants in Cohort 6 received an intravenous 8.0 mg/kg dose of DS-8201a (FL-DP1).
- Dose Expansion: HER2-positive Breast Cancer, 5.4 mg/kg: Participants with HER2-overexpressing breast cancer received an intravenous 5.4 mg/kg dose of DS-8201a (FL-DP1).
- Dose Expansion: HER2-positive Breast Cancer, 6.4 mg/kg: Participants with HER2-overexpressing breast cancer received an intravenous 6.4 mg/kg dose of DS-8201a (FL-DP1).
- Dose Expansion: HER2-low Expressing Breast Cancer, 5.4 mg/kg: Participants with HER2-low expressing breast cancer received an intravenous 5.4 mg/kg dose of DS-8201a (FL-DP1).
- Dose Expansion: HER2-low Expressing Breast Cancer, 6.4 mg/kg: Participants with HER2-low expressing breast cancer received an intravenous 6.4 mg/kg dose of DS-8201a (FL-DP1).
- Dose Expansion: HER2-overexpressing Gastric or GEJ, 5.4 mg/kg: Participants with HER2-overexpressing gastric or gastroesophageal junction (GEJ) adenocarcinoma received an intravenous 5.4 mg/kg dose of DS-8201a (FL-DP1).
- Dose Expansion: HER2-overexpressing Gastric or GEJ, 6.4 mg/kg: Participants with HER2-overexpressing gastric or gastroesophageal junction (GEJ) adenocarcinoma received an intravenous 6.4 mg/kg dose of DS-8201a (FL-DP1).
- Dose Expansion: HER2-expressing NSCLC Tumors: Participants with HER2-expressing NSCLC tumors received an intravenous 6.4 mg/kg dose of DS-8201a (FL-DP1).
- Dose Expansion: HER2-expressing Colorectal Tumors: Participants with HER2-expressing colorectal tumors received an intravenous 6.4 mg/kg dose of DS-8201a (FL-DP1).
- Dose Expansion: HER2-expressing Other Solid Tumors: Participants with any other HER2-expressing solid tumor other than breast or gastric or any tumor with HER2 mutation received an intravenous 6.4 mg/kg dose of DS-8201a (FL-DP1).
Period: Dose Escalation
Arm/Group | Dose Escalation: Cohort 1, 0.8 mg/kg | Dose Escalation: Cohort 2, 1.6 mg/kg | Dose Escalation: Cohort 3, 3.2 mg/kg | Dose Escalation: Cohort 4, 5.4 mg/kg | Dose Escalation: Cohort 5, 6.4 mg/kg | Dose Escalation: Cohort 6, 8.0 mg/kg | Dose Expansion: HER2-positive Breast Cancer, 5.4 mg/kg | Dose Expansion: HER2-positive Breast Cancer, 6.4 mg/kg | Dose Expansion: HER2-low Expressing Breast Cancer, 5.4 mg/kg | Dose Expansion: HER2-low Expressing Breast Cancer, 6.4 mg/kg | Dose Expansion: HER2-overexpressing Gastric or GEJ, 5.4 mg/kg | Dose Expansion: HER2-overexpressing Gastric or GEJ, 6.4 mg/kg | Dose Expansion: HER2-expressing NSCLC Tumors | Dose Expansion: HER2-expressing Colorectal Tumors | Dose Expansion: HER2-expressing Other Solid Tumors
Started | 3 | 3 | 3 | 6 | 6 | 6 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Completed (Data from Ongoing and Discontinued participants are presented as of data cutoff on 01 February 2019) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 3 | 3 | 3 | 6 | 6 | 6 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Progressive disease per RECIST | 2 | 3 | 3 | 3 | 3 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Ongoing | 1 | 0 | 0 | 2 | 2 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 0 | 0 | 0 | 1 | 1 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Dose Expansion
Arm/Group | Dose Escalation: Cohort 1, 0.8 mg/kg | Dose Escalation: Cohort 2, 1.6 mg/kg | Dose Escalation: Cohort 3, 3.2 mg/kg | Dose Escalation: Cohort 4, 5.4 mg/kg | Dose Escalation: Cohort 5, 6.4 mg/kg | Dose Escalation: Cohort 6, 8.0 mg/kg | Dose Expansion: HER2-positive Breast Cancer, 5.4 mg/kg | Dose Expansion: HER2-positive Breast Cancer, 6.4 mg/kg | Dose Expansion: HER2-low Expressing Breast Cancer, 5.4 mg/kg | Dose Expansion: HER2-low Expressing Breast Cancer, 6.4 mg/kg | Dose Expansion: HER2-overexpressing Gastric or GEJ, 5.4 mg/kg | Dose Expansion: HER2-overexpressing Gastric or GEJ, 6.4 mg/kg | Dose Expansion: HER2-expressing NSCLC Tumors | Dose Expansion: HER2-expressing Colorectal Tumors | Dose Expansion: HER2-expressing Other Solid Tumors
Started (Only the Dose Expansion Phase is being presented.) | 0 | 0 | 0 | 0 | 0 | 0 | 49 | 62 | 20 | 33 | 17 | 24 | 18 | 20 | 22
Enrolled, But Not Dosed | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Completed (Data from Ongoing and Discontinued participants are presented as of data cutoff on 01 February 2019.) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 49 | 62 | 20 | 33 | 17 | 24 | 18 | 20 | 22
Not completed — Progressive disease per RECIST | 0 | 0 | 0 | 0 | 0 | 0 | 19 | 17 | 8 | 16 | 13 | 19 | 10 | 13 | 11
Not completed — Clinical progression | 0 | 0 | 0 | 0 | 0 | 0 | 5 | 12 | 0 | 3 | 2 | 0 | 1 | 3 | 1
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 0 | 0 | 9 | 22 | 0 | 11 | 0 | 5 | 2 | 2 | 1
Not completed — Ongoing | 0 | 0 | 0 | 0 | 0 | 0 | 9 | 10 | 11 | 3 | 0 | 0 | 4 | 0 | 6
Not completed — Death | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 1
Not completed — Other | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Did not receive treatment | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Demographic and baseline characteristics were assessed in the Enrolled Analysis Set (Dose Escalation, n=27; Dose Expansion, n=265).
Groups:
- Total: Total of all reporting groups
Arm/Group | Dose Escalation: Cohort 1, 0.8 mg/kg | Dose Escalation: Cohort 2, 1.6 mg/kg | Dose Escalation: Cohort 3, 3.2 mg/kg | Dose Escalation: Cohort 4, 5.4 mg/kg | Dose Escalation: Cohort 5, 6.4 mg/kg | Dose Escalation: Cohort 6, 8.0 mg/kg | Dose Expansion: HER2-positive Breast Cancer, 5.4 mg/kg | Dose Expansion: HER2-positive Breast Cancer, 6.4 mg/kg | Dose Expansion: HER2-low Expressing Breast Cancer, 5.4 mg/kg | Dose Expansion: HER2-low Expressing Breast Cancer, 6.4 mg/kg | Dose Expansion: HER2-overexpressing Gastric or GEJ, 5.4 mg/kg | Dose Expansion: HER2-overexpressing Gastric or GEJ, 6.4 mg/kg | Dose Expansion: HER2-expressing NSCLC Tumors | Dose Expansion: HER2-expressing Colorectal Tumors | Dose Expansion: HER2-expressing Other Solid Tumors | Total
Number analyzed (Participants) | 3 | 3 | 3 | 6 | 6 | 6 | 49 | 62 | 20 | 33 | 17 | 24 | 18 | 20 | 22 | 292
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 2 | 1 | 2 | 2 | 4 | 2 | 33 | 48 | 14 | 25 | 6 | 8 | 12 | 16 | 16 | 191
  >=65 years | 1 | 2 | 1 | 4 | 2 | 4 | 16 | 14 | 6 | 8 | 11 | 16 | 6 | 4 | 6 | 101
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.3 (7.09) | 66.3 (4.73) | 48.3 (14.57) | 66.8 (14.82) | 58.2 (10.40) | 66.2 (10.67) | 56.2 (12.11) | 54.9 (10.28) | 57.8 (9.68) | 56.3 (10.97) | 64.2 (11.00) | 66.2 (8.55) | 57.4 (15.29) | 59.5 (9.90) | 58.5 (10.16) | 58.1 (11.39)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 3 | 3 | 6 | 6 | 5 | 48 | 62 | 20 | 33 | 5 | 4 | 13 | 9 | 9 | 229
  Male | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 12 | 20 | 5 | 11 | 13 | 63
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Asian | 3 | 3 | 3 | 6 | 6 | 3 | 25 | 40 | 6 | 23 | 11 | 24 | 9 | 17 | 14 | 193
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Black or African American | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 2 | 1 | 1 | 0 | 0 | 1 | 0 | 0 | 8
  White | 0 | 0 | 0 | 0 | 0 | 3 | 19 | 19 | 12 | 7 | 5 | 0 | 8 | 3 | 7 | 83
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 2
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 4
Region of Enrollment [Number; unit: participants]
  United States | 0 | 0 | 0 | 0 | 0 | 3 | 30 | 25 | 16 | 11 | 5 | 0 | 10 | 3 | 9 | 112
  Japan | 3 | 3 | 3 | 6 | 6 | 3 | 19 | 37 | 4 | 22 | 12 | 24 | 8 | 17 | 13 | 180

OUTCOME MEASURES:

1. Primary Outcome: Objective Response Rate (ORR) Following Treatment With DS-8201a in Participants With Advanced Solid Malignant Tumors (Dose Escalation and Dose Expansion Phases)
Description: Objective response rate (ORR) by independent central review was defined as the proportion of participants who achieve either complete response [CR] or partial response [PR] per Response Evaluation Criteria in Solid Tumors (RECIST) v1.1. CR was defined as a disappearance of all target lesions and PR was defined as at least a 30% decrease in the sum of diameters of target lesions. HER2-positive other solid tumors included participants with salivary/submandibular/parotid gland (8 participants), breast with HER2-mutation (2 participants), endometrial (2 participants), esophageal (2 participants), Paget's disease (2 participants), cholangiocarcinoma (1 participant), extraskeletal myxoide chondrosarcoma (1 participant), gallbladder (1 participant), pancreatic (1 participant), small intestine (1 participant), uterine cervix (1 participant) and HER2-low gastric/GEJ (1 participant who received 5.4 mg/kg) cancer.
Time Frame: From 6 months postdose of last participant up to 3 years 5 months
Population: ORR was assessed among participants in the Intent-to-Treat Analysis Set.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Dose Expansion: HER2-overexpressing Gastric or GEJ, 5.4 mg/kg; Dose Expansion: HER2-overexpressing Gastric or GEJ, 6.4 mg/kg: Participants with HER2-overexpressing gastric or gastroesophageal junction (GEJ) adenocarcinoma received an intravenous 6.4 mg/kg dose of DS-8201a (FL-DP1).
Arm/Group | Dose Escalation: Cohort 1, 0.8 mg/kg | Dose Escalation: Cohort 2, 1.6 mg/kg | Dose Escalation: Cohort 3, 3.2 mg/kg | Dose Escalation: Cohort 4, 5.4 mg/kg | Dose Escalation: Cohort 5, 6.4 mg/kg | Dose Escalation: Cohort 6, 8.0 mg/kg | Dose Expansion: HER2-positive Breast Cancer, 5.4 mg/kg | Dose Expansion: HER2-positive Breast Cancer, 6.4 mg/kg | Dose Expansion: HER2-low Expressing Breast Cancer, 5.4 mg/kg | Dose Expansion: HER2-low Expressing Breast Cancer, 6.4 mg/kg | Dose Expansion: HER2-overexpressing Gastric or GEJ, 5.4 mg/kg | Dose Expansion: HER2-overexpressing Gastric or GEJ, 6.4 mg/kg | Dose Expansion: HER2-expressing NSCLC Tumors | Dose Expansion: HER2-expressing Colorectal Tumors | Dose Expansion: HER2-expressing Other Solid Tumors
Number analyzed (Participants) | 3 | 3 | 3 | 6 | 6 | 6 | 51 | 67 | 21 | 33 | 19 | 25 | 18 | 20 | 23
percentage of participants | 0 [0 to 70.8] | 33.3 [0.8 to 90.6] | 0 [0 to 70.8] | 83.3 [35.9 to 99.6] | 33.3 [4.3 to 77.7] | 50.0 [11.8 to 88.2] | 51.0 [36.6 to 65.2] | 53.7 [41.1 to 66.0] | 33.3 [14.6 to 57.0] | 39.4 [22.9 to 57.9] | 26.3 [9.1 to 51.2] | 32.0 [14.9 to 53.5] | 55.6 [30.8 to 78.5] | 5.0 [0.1 to 24.9] | 30.4 [13.2 to 52.9]

2. Secondary Outcome: Disease Control Rate (DCR) Following Treatment With DS-8201a in Participants With Advanced Solid Malignant Tumors (Dose Escalation and Dose Expansion Phases)
Description: Disease control rate (DCR) by independent central review was calculated as the proportion of participants demonstrating complete response (CR), partial response (PR), or stable disease (SD) for a minimum of 6 weeks (±1week) from the first dosing date. CR was defined as a disappearance of all target lesions, PR as at least a 30% decrease in the sum of diameters of target lesions, and stable disease (SD) was defined as neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for progressive disease (PD; at least a 20% increase in the sum of diameters of target lesions. HER2-positive other solid tumors included 8 participants with salivary/submandibular/parotid gland, 2 breast with HER2-mutation, 2 endometrial, 2 esophageal, 2 Paget's disease, 1 cholangiocarcinoma, 1 extraskeletal myxoide chondrosarcoma, 1 gallbladder, 1 pancreatic, 1 small intestine, 1 uterine cervix, and 1 participant who received 5.4 mg/kg with HER2-low gastric/GEJ cancer.
Time Frame: From 6 months postdose of last participant up to 3 years 5 months
Population: DCR was assessed in the Intent-to-Treat Analysis Set.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Dose Escalation: Cohort 1, 0.8 mg/kg | Dose Escalation: Cohort 2, 1.6 mg/kg | Dose Escalation: Cohort 3, 3.2 mg/kg | Dose Escalation: Cohort 4, 5.4 mg/kg | Dose Escalation: Cohort 5, 6.4 mg/kg | Dose Escalation: Cohort 6, 8.0 mg/kg | Dose Expansion: HER2-positive Breast Cancer, 5.4 mg/kg | Dose Expansion: HER2-positive Breast Cancer, 6.4 mg/kg | Dose Expansion: HER2-low Expressing Breast Cancer, 5.4 mg/kg | Dose Expansion: HER2-low Expressing Breast Cancer, 6.4 mg/kg | Dose Expansion: HER2-overexpressing Gastric or GEJ, 5.4 mg/kg | Dose Expansion: HER2-overexpressing Gastric or GEJ, 6.4 mg/kg | Dose Expansion: HER2-expressing NSCLC Tumors | Dose Expansion: HER2-expressing Colorectal Tumors | Dose Expansion: HER2-expressing Other Solid Tumors
Number analyzed (Participants) | 3 | 3 | 3 | 6 | 6 | 6 | 51 | 67 | 21 | 33 | 19 | 25 | 18 | 20 | 23
percentage of participants | 100.0 [29.2 to 100.0] | 100.0 [29.2 to 100.0] | 66.7 [9.4 to 99.2] | 100.0 [54.1 to 100.0] | 100.0 [54.1 to 100.0] | 100.0 [54.1 to 100.0] | 88.2 [76.1 to 95.6] | 95.5 [87.5 to 99.1] | 85.7 [63.7 to 97.0] | 87.9 [71.8 to 96.6] | 78.9 [54.4 to 93.9] | 88.0 [68.8 to 97.5] | 83.3 [58.6 to 96.4] | 80.0 [56.3 to 94.3] | 82.6 [61.2 to 95.0]

3. Secondary Outcome: Best Overall Response Following Treatment With DS-8201a in Participants With Advanced Solid Malignant Tumors (Dose Escalation and Dose Expansion Phases)
Description: Best overall response by independent central review was defined as the proportion of participants who achieved either complete response [CR], partial response [PR], stable disease (SD), progressive disease (PD), or were non-evaluable (NE) as per RECIST v1.1. CR was defined as a disappearance of all target lesions, PR at least a 30% decrease in the sum of diameters of target lesions, and SD as neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD defined as at least a 20% increase in the sum of diameters of target lesions. HER2-positive other solid tumors included 8 participants with salivary/submandibular/parotid gland, 2 breast with HER2-mutation, 2 endometrial, 2 esophageal, 2 Paget's disease, 1 cholangiocarcinoma, 1 extraskeletal myxoide chondrosarcoma, 1 gallbladder, 1 pancreatic, 1 small intestine, 1 uterine cervix, and 1 participant who received 5.4 mg/kg with HER2-low gastric/GEJ cancer.
Time Frame: From 6 months postdose of last participant up to 3 years 5 months
Population: Best overall response was assessed in the Intent-to-Treat Analysis Set.
Measure: Count of Participants; unit: Participants
Arm/Group | Dose Escalation: Cohort 1, 0.8 mg/kg | Dose Escalation: Cohort 2, 1.6 mg/kg | Dose Escalation: Cohort 3, 3.2 mg/kg | Dose Escalation: Cohort 4, 5.4 mg/kg | Dose Escalation: Cohort 5, 6.4 mg/kg | Dose Escalation: Cohort 6, 8.0 mg/kg | Dose Expansion: HER2-positive Breast Cancer, 5.4 mg/kg | Dose Expansion: HER2-positive Breast Cancer, 6.4 mg/kg | Dose Expansion: HER2-low Expressing Breast Cancer, 5.4 mg/kg | Dose Expansion: HER2-low Expressing Breast Cancer, 6.4 mg/kg | Dose Expansion: HER2-overexpressing Gastric or GEJ, 5.4 mg/kg | Dose Expansion: HER2-overexpressing Gastric or GEJ, 6.4 mg/kg | Dose Expansion: HER2-expressing NSCLC Tumors | Dose Expansion: HER2-expressing Colorectal Tumors | Dose Expansion: HER2-expressing Other Solid Tumors
Number analyzed (Participants) | 3 | 3 | 3 | 6 | 6 | 6 | 51 | 67 | 21 | 33 | 19 | 25 | 18 | 20 | 23
Participants
  Complete response | 0 | 0 | 0 | 1 | 1 | 0 | 2 | 8 | 0 | 0 | 0 | 1 | 0 | 0 | 2
  Partial response | 0 | 1 | 0 | 4 | 1 | 3 | 24 | 28 | 7 | 13 | 5 | 7 | 10 | 1 | 5
  Stable disease | 3 | 2 | 2 | 1 | 4 | 3 | 19 | 28 | 11 | 16 | 10 | 14 | 5 | 15 | 12
  Progressive disease | 0 | 0 | 1 | 0 | 0 | 0 | 4 | 1 | 3 | 3 | 4 | 3 | 2 | 2 | 3
  Non-evaluable | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 2 | 0 | 1 | 0 | 0 | 1 | 2 | 1

4. Secondary Outcome: Duration of Response (DoR) Following Treatment With DS-8201a in Participants With Advanced Solid Malignant Tumors (Dose Expansion Phases)
Description: Duration of response (DoR) by independent central review was defined as the time between the date of the first complete response (CR) or partial response (PR) until the date of the first documentation of progressive disease (PD) or death due to any cause. CR was defined as a disappearance of all target lesions, PR as at least a 30% decrease in the sum of diameters of target lesions, and PD as at least a 20% increase in the sum of diameters of target lesions. HER2-positive other solid tumors included participants with salivary/submandibular/parotid gland (8 participants), breast with HER2-mutation (2 participants), endometrial (2 participants), esophageal (2 participants), Paget's disease (2 participants), cholangiocarcinoma (1 participant), extraskeletal myxoide chondrosarcoma (1 participant), gallbladder (1 participant), pancreatic (1 participant), small intestine (1 participant), uterine cervix (1 participant) and HER2-low gastric/GEJ (1 participant who received 5.4 mg/kg) cancer.
Time Frame: From 6 months postdose of last participant up to 3 years 5 months
Population: DoR was assessed among participants who achieved a CR or PR in the Intent-to-Treat Analysis Set.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Dose Expansion: HER2-positive Breast Cancer, 5.4 mg/kg | Dose Expansion: HER2-positive Breast Cancer, 6.4 mg/kg | Dose Expansion: HER2-low Expressing Breast Cancer, 5.4 mg/kg | Dose Expansion: HER2-low Expressing Breast Cancer, 6.4 mg/kg | Dose Expansion: HER2-overexpressing Gastric or GEJ, 5.4 mg/kg | Dose Expansion: HER2-overexpressing Gastric or GEJ, 6.4 mg/kg | Dose Expansion: HER2-expressing NSCLC Tumors | Dose Expansion: HER2-expressing Colorectal Tumors | Dose Expansion: HER2-expressing Other Solid Tumors
Number analyzed (Participants) | 51 | 67 | 21 | 33 | 19 | 25 | 18 | 20 | 23
months | 12.7 [6.7 to NA] — Missing upper bound is related to right-censored data. Last time point censored and estimate is essentially infinity, therefore it is NA. | 13.6 [7.3 to NA] — Missing upper bound is related to right-censored data. Last time point censored and estimate is essentially infinity, therefore it is NA. | NA [NA to NA] — Lack of a median value is due to less than 50% of the participants experiencing the event. In a Kaplan-Meier analysis, the curve would never fall below the 50% mark, and would continue to the largest observed censored time value. | 10.4 [3.4 to NA] — Missing upper bound is related to right-censored data. Last time point censored and estimate is essentially infinity, therefore it is NA. | 5.6 [2.9 to NA] — Missing upper bound is related to right-censored data. Last time point censored and estimate is essentially infinity, therefore it is NA. | 6.9 [3.5 to NA] — Missing upper bound is related to right-censored data. Last time point censored and estimate is essentially infinity, therefore it is NA. | 10.7 [6.9 to 11.5] | 13.4 [NA to NA] — Missing upper bound is related to right-censored data. Last time point censored and estimate is essentially infinity, therefore it is NA. | NA [3.0 to NA] — Median and 95% confidence interval were not calculable due to insufficient number of participants with events.

5. Secondary Outcome: Time to Response (TTR) Following Treatment With DS-8201a in Participants With Advanced Solid Malignant Tumors (Dose Expansion Phases)
Description: Time to response (TTR) by independent central review was defined as the time interval between the date of registration until the date at which the criteria were first met for complete response (CR) or partial response (PR). Only participants who achieved CR or PR were included in the TTR analysis. CR was defined as a disappearance of all target lesions and PR was defined as at least a 30% decrease in the sum of diameters of target lesions. HER2-positive other solid tumors included participants with salivary/submandibular/parotid gland (8 participants), breast with HER2-mutation (2 participants), endometrial (2 participants), esophageal (2 participants), Paget's disease (2 participants), cholangiocarcinoma (1 participant), extraskeletal myxoide chondrosarcoma (1 participant), gallbladder (1 participant), pancreatic (1 participant), small intestine (1 participant), uterine cervix (1 participant) and HER2-low gastric/GEJ (1 participant who received 5.4 mg/kg) cancer.
Time Frame: From 6 months postdose of last participant up to 3 years 5 months
Population: Time to response was assessed among participants who achieved CR or PR in the Intent-to-Treat Analysis Set.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Dose Expansion: HER2-positive Breast Cancer, 5.4 mg/kg | Dose Expansion: HER2-positive Breast Cancer, 6.4 mg/kg | Dose Expansion: HER2-low Expressing Breast Cancer, 5.4 mg/kg | Dose Expansion: HER2-low Expressing Breast Cancer, 6.4 mg/kg | Dose Expansion: HER2-overexpressing Gastric or GEJ, 5.4 mg/kg | Dose Expansion: HER2-overexpressing Gastric or GEJ, 6.4 mg/kg | Dose Expansion: HER2-expressing NSCLC Tumors | Dose Expansion: HER2-expressing Colorectal Tumors | Dose Expansion: HER2-expressing Other Solid Tumors
Number analyzed (Participants) | 51 | 67 | 21 | 33 | 19 | 25 | 18 | 20 | 23
months | 2.7 [1.5 to 2.9] | 2.8 [1.4 to 2.9] | 2.6 [1.2 to 4.2] | 2.7 [1.2 to 3.1] | 1.6 [1.2 to 3.1] | 2.2 [1.4 to 2.9] | 1.4 [1.2 to 2.8] | 3.0 [NA to NA] — The 95% confidence interval was not calculable due to insufficient number of participants with events. | 1.6 [1.2 to 2.9]

6. Secondary Outcome: Progression-free Survival Following Treatment With DS-8201a in Participants With Advanced Solid Malignant Tumors (Dose Expansion Phases)
Description: Progression-free survival (PFS) by independent central review was defined as the time from the date of enrollment to the earlier of the dates of the first objective documentation of disease progression (as per RECIST v1.1) or death due to any cause. Progressive disease was defined as at least a 20% increase in the sum of diameters of target lesions. HER2-positive other solid tumors included participants with salivary/submandibular/parotid gland (8 participants), breast with HER2-mutation (2 participants), endometrial (2 participants), esophageal (2 participants), Paget's disease (2 participants), cholangiocarcinoma (1 participant), extraskeletal myxoide chondrosarcoma (1 participant), gallbladder (1 participant), pancreatic (1 participant), small intestine (1 participant), uterine cervix (1 participant) and HER2-low gastric/GEJ (1 participant who received 5.4 mg/kg) cancer.
Time Frame: From 6 months postdose of last participant up to 3 years 5 months
Population: PFS was assessed in the Intent-to-Treat Analysis Set.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Dose Expansion: HER2-positive Breast Cancer, 5.4 mg/kg | Dose Expansion: HER2-positive Breast Cancer, 6.4 mg/kg | Dose Expansion: HER2-low Expressing Breast Cancer, 5.4 mg/kg | Dose Expansion: HER2-low Expressing Breast Cancer, 6.4 mg/kg | Dose Expansion: HER2-overexpressing Gastric or GEJ, 5.4 mg/kg | Dose Expansion: HER2-overexpressing Gastric or GEJ, 6.4 mg/kg | Dose Expansion: HER2-expressing NSCLC Tumors | Dose Expansion: HER2-expressing Colorectal Tumors | Dose Expansion: HER2-expressing Other Solid Tumors
Number analyzed (Participants) | 51 | 67 | 21 | 33 | 19 | 25 | 18 | 20 | 23
months | 13.7 [8.5 to 19.6] | 14.1 [8.5 to NA] — Missing upper bound is related to right-censored data. Last time point censored and estimate is essentially infinity, therefore it is NA. | NA [2.7 to NA] — Median and 95% confidence interval were not calculable due to insufficient number of participants with events. | 11.1 [5.0 to NA] — Missing upper bound is related to right-censored data. Last time point censored and estimate is essentially infinity, therefore it is NA. | 4.3 [2.6 to 8.6] | 8.2 [4.2 to 11.0] | 11.3 [7.2 to 14.3] | 4.0 [2.7 to 5.6] | 11.0 [2.8 to NA] — Missing upper bound is related to right-censored data. Last time point censored and estimate is essentially infinity, therefore it is NA.

7. Secondary Outcome: Overall Survival Among Participants With Advanced Solid Malignant Tumors (Dose Expansion Phases)
Description: Overall survival (OS) by independent central review was defined as the time interval from the date of enrollment to the date of death from any cause. HER2-positive other solid tumors included participants with salivary/submandibular/parotid gland (8 participants), breast with HER2-mutation (2 participants), endometrial (2 participants), esophageal (2 participants), Paget's disease (2 participants), cholangiocarcinoma (1 participant), extraskeletal myxoide chondrosarcoma (1 participant), gallbladder (1 participant), pancreatic (1 participant), small intestine (1 participant), uterine cervix (1 participant) and HER2-low gastric/GEJ (1 participant who received 5.4 mg/kg) cancer.
Time Frame: From 6 months postdose of last participant up to 3 years 5 months
Population: OS was assessed in the Intent-to-Treat Analysis Set.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Dose Expansion: HER2-positive Breast Cancer, 5.4 mg/kg | Dose Expansion: HER2-positive Breast Cancer, 6.4 mg/kg | Dose Expansion: HER2-low Expressing Breast Cancer, 5.4 mg/kg | Dose Expansion: HER2-low Expressing Breast Cancer, 6.4 mg/kg | Dose Expansion: HER2-overexpressing Gastric or GEJ, 5.4 mg/kg | Dose Expansion: HER2-overexpressing Gastric or GEJ, 6.4 mg/kg | Dose Expansion: HER2-expressing NSCLC Tumors | Dose Expansion: HER2-expressing Colorectal Tumors | Dose Expansion: HER2-expressing Other Solid Tumors
Number analyzed (Participants) | 51 | 67 | 21 | 33 | 19 | 25 | 18 | 20 | 23
months | NA [NA to NA] — Lack of median value is due to less than 50% of the participants experiencing the event. In a Kaplan-Meier analysis, the curve would never fall below the 50% mark, and would continue to the largest observed censored time value. | NA [26.4 to NA] — Median and 95% confidence interval were not calculable due to insufficient number of participants with events. | NA [NA to NA] — Lack of median value is due to less than 50% of the participants experiencing the event. In a Kaplan-Meier analysis, the curve would never fall below the 50% mark, and would continue to the largest observed censored time value. | 19.7 [12.5 to 29.4] | 18.9 [5.7 to NA] — Missing upper bound is related to right-censored data. Last time point censored and estimate is essentially infinity, therefore it is NA. | 26.2 [10.0 to NA] — Missing upper bound is related to right-censored data. Last time point censored and estimate is essentially infinity, therefore it is NA. | NA [17.3 to NA] — Median and 95% confidence interval were not calculable due to insufficient number of participants with events. | 15.6 [4.8 to NA] — Missing upper bound is related to right-censored data. Last time point censored and estimate is essentially infinity, therefore it is NA. | 23.4 [9.7 to NA] — Missing upper bound is related to right-censored data. Last time point censored and estimate is essentially infinity, therefore it is NA.

8. Secondary Outcome: Pharmacokinetic (PK) Analysis: Area Under the Concentration Versus Time Curve (AUC) of Serum DS-8201a Following First Dose
Description: The serum PK parameters of DS-8201a and its analytes for area under the concentration-versus-time curve from time 0 to the last quantifiable concentration as calculated by the linear-up log-down trapezoidal method (AUClast) and AUC from time 0 to infinity (AUCinf) elimination rate constant associated with the terminal phase were estimated using standard non-compartmental methods.
Time Frame: Post first dose up to Day 147
Population: Pharmacokinetic parameters were assessed in the Pharmacokinetic Analysis Set.
Measure: Mean (Standard Deviation); unit: ug*d/mL
Groups:
- Dose Expansion: HER2-expressing Breast Cancer: Japan only: Participants with HER2-expressing breast cancer received an intravenous 6.4 mg/kg dose of DS-8201a (FL-DP2).
Arm/Group | Dose Escalation: Cohort 1, 0.8 mg/kg | Dose Escalation: Cohort 2, 1.6 mg/kg | Dose Escalation: Cohort 3, 3.2 mg/kg | Dose Escalation: Cohort 4, 5.4 mg/kg | Dose Escalation: Cohort 5, 6.4 mg/kg | Dose Escalation: Cohort 6, 8.0 mg/kg | Dose Expansion: HER2-positive Breast Cancer, 5.4 mg/kg | Dose Expansion: HER2-positive Breast Cancer, 6.4 mg/kg | Dose Expansion: HER2-low Expressing Breast Cancer, 5.4 mg/kg | Dose Expansion: HER2-low Expressing Breast Cancer, 6.4 mg/kg | Dose Expansion: HER2-overexpressing Gastric or GEJ, 5.4 mg/kg | Dose Expansion: HER2-overexpressing Gastric or GEJ, 6.4 mg/kg | Dose Expansion: HER2-expressing Other Solid Tumors | Dose Expansion: HER2-expressing Breast Cancer
Number analyzed (Participants) | 3 | 3 | 3 | 6 | 6 | 5 | 48 | 50 | 20 | 19 | 17 | 23 | 58 | 21
ug*d/mL
  AUClast | 51.7 (13.1) | 116 (58.7) | 325 (142) | 544 (165) | 901 (155) | 996 (229) | 559 (178) | 785 (228) | 581 (180) | 693 (178) | 542 (163) | 507 (126) | 631 (184) | 693 (102)
  AUCinfinity: number analyzed (Participants) | 3 | 3 | 3 | 6 | 6 | 5 | 48 | 49 | 19 | 17 | 17 | 22 | 58 | 21
  AUCinfinity | 55.0 (11.9) | 121 (58.9) | 340 (150) | 590 (186) | 1030 (209) | 1100 (259) | 602 (203) | 848 (243) | 589 (145) | 762 (205) | 596 (183) | 563 (151) | 683 (209) | 753 (118)

9. Secondary Outcome: Pharmacokinetic Analysis: Maximum (Peak) Observed Serum Concentration (Cmax) of Serum DS-8201a Following First Dose
Description: The serum PK parameters Maximum (peak) Observed serum concentration of DS-8201a and its analytes were estimated using standard non-compartmental method.
Time Frame: Post first dose up to Day 147
Population: Pharmacokinetic parameters were assessed in the Pharmacokinetic Analysis Set.
Measure: Mean (Standard Deviation); unit: ug/mL
Arm/Group | Dose Escalation: Cohort 1, 0.8 mg/kg | Dose Escalation: Cohort 2, 1.6 mg/kg | Dose Escalation: Cohort 3, 3.2 mg/kg | Dose Escalation: Cohort 4, 5.4 mg/kg | Dose Escalation: Cohort 5, 6.4 mg/kg | Dose Escalation: Cohort 6, 8.0 mg/kg | Dose Expansion: HER2-positive Breast Cancer, 5.4 mg/kg | Dose Expansion: HER2-positive Breast Cancer, 6.4 mg/kg | Dose Expansion: HER2-low Expressing Breast Cancer, 5.4 mg/kg | Dose Expansion: HER2-low Expressing Breast Cancer, 6.4 mg/kg | Dose Expansion: HER2-overexpressing Gastric or GEJ, 5.4 mg/kg | Dose Expansion: HER2-overexpressing Gastric or GEJ, 6.4 mg/kg | Dose Expansion: HER2-expressing Other Solid Tumors | Dose Expansion: HER2-expressing Breast Cancer
Number analyzed (Participants) | 3 | 3 | 3 | 6 | 6 | 5 | 48 | 50 | 20 | 19 | 17 | 23 | 59 | 21
ug/mL | 22.9 (3.76) | 36.2 (4.98) | 78.2 (16.1) | 127 (17.2) | 181 (33.1) | 221 (41.0) | 126 (37.7) | 170 (53.6) | 133 (18.3) | 155 (33.2) | 113 (30.0) | 116 (21.1) | 150 (30.3) | 155 (21.4)

10. Secondary Outcome: Pharmacokinetic Analysis: Time of Maximum Plasma Concentration (Tmax) of Serum DS-8201a Following First Dose
Description: The serum PK parameters of Time of maximum plasma concentration (Tmax) for DS-8201a and its analytes were estimated using standard non-compartmental methods.
Time Frame: Post first dose up to Day 147
Population: Pharmacokinetic parameters were assessed in the Pharmacokinetic Analysis Set.
Measure: Median (Full Range); unit: hours
Arm/Group | Dose Escalation: Cohort 1, 0.8 mg/kg | Dose Escalation: Cohort 2, 1.6 mg/kg | Dose Escalation: Cohort 3, 3.2 mg/kg | Dose Escalation: Cohort 4, 5.4 mg/kg | Dose Escalation: Cohort 5, 6.4 mg/kg | Dose Escalation: Cohort 6, 8.0 mg/kg | Dose Expansion: HER2-positive Breast Cancer, 5.4 mg/kg | Dose Expansion: HER2-positive Breast Cancer, 6.4 mg/kg | Dose Expansion: HER2-low Expressing Breast Cancer, 5.4 mg/kg | Dose Expansion: HER2-low Expressing Breast Cancer, 6.4 mg/kg | Dose Expansion: HER2-overexpressing Gastric or GEJ, 5.4 mg/kg | Dose Expansion: HER2-overexpressing Gastric or GEJ, 6.4 mg/kg | Dose Expansion: HER2-expressing Other Solid Tumors | Dose Expansion: HER2-expressing Breast Cancer
Number analyzed (Participants) | 3 | 3 | 3 | 6 | 6 | 5 | 48 | 50 | 20 | 19 | 17 | 23 | 59 | 21
hours | 1.95 [1.62 to 1.98] | 4.03 [1.87 to 4.08] | 4.12 [1.95 to 6.88] | 2.02 [1.87 to 2.07] | 2.06 [1.50 to 3.97] | 1.97 [1.70 to 6.80] | 2.00 [1.50 to 6.85] | 2.08 [1.53 to 7.05] | 2.16 [1.50 to 7.07] | 2.00 [1.50 to 6.67] | 2.03 [1.58 to 4.08] | 1.95 [1.53 to 7.00] | 2.02 [1.50 to 7.20] | 2.05 [1.62 to 7.23]

11. Secondary Outcome: Pharmacokinetic Analysis: Terminal Elimination Half-life (t1/2) of Serum DS-8201a Following First Dose
Description: The serum PK parameters of Terminal elimination half-life for DS-8201a and its analytes was estimated using standard non-compartmental methods.
Time Frame: Post first dose up to Day 147
Population: Pharmacokinetic parameters were assessed in the Pharmacokinetic Analysis Set.
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Dose Escalation: Cohort 1, 0.8 mg/kg | Dose Escalation: Cohort 2, 1.6 mg/kg | Dose Escalation: Cohort 3, 3.2 mg/kg | Dose Escalation: Cohort 4, 5.4 mg/kg | Dose Escalation: Cohort 5, 6.4 mg/kg | Dose Escalation: Cohort 6, 8.0 mg/kg | Dose Expansion: HER2-positive Breast Cancer, 5.4 mg/kg | Dose Expansion: HER2-positive Breast Cancer, 6.4 mg/kg | Dose Expansion: HER2-low Expressing Breast Cancer, 5.4 mg/kg | Dose Expansion: HER2-low Expressing Breast Cancer, 6.4 mg/kg | Dose Expansion: HER2-overexpressing Gastric or GEJ, 5.4 mg/kg | Dose Expansion: HER2-overexpressing Gastric or GEJ, 6.4 mg/kg | Dose Expansion: HER2-expressing Other Solid Tumors | Dose Expansion: HER2-expressing Breast Cancer
Number analyzed (Participants) | 3 | 3 | 3 | 6 | 6 | 5 | 48 | 49 | 19 | 17 | 17 | 22 | 58 | 21
days | 2.18 (0.671) | 3.07 (1.22) | 4.23 (1.24) | 6.03 (0.603) | 7.33 (1.64) | 6.44 (0.793) | 5.52 (1.23) | 6.00 (1.22) | 5.28 (1.49) | 5.79 (1.01) | 6.18 (1.18) | 5.90 (1.57) | 5.61 (1.29) | 5.46 (1.02)

12. Secondary Outcome: Overview of Treatment-emergent Adverse Events
Description: Treatment-emergent adverse events were graded by Common Terminology Criteria for Adverse Events, v4.03.
Time Frame: Baseline up to 28 days after the last dose of study drug, up to 3 years 5 months
Population: Safety events were assessed in the Safety Analysis Set. It was prespecified in the protocol that single patients with unique tumor types would be combined into 1 group for the safety analysis. For the safety overview, TEAEs for HER2-expressing NSCLC, Colorectal, and Other Solid Tumors (excluding 1 HER2-low gastric cancer subject who received 5.4 mg/kg) were combined and reported together.
Measure: Count of Participants; unit: Participants
Arm/Group | Dose Escalation: Cohort 1, 0.8 mg/kg | Dose Escalation: Cohort 2, 1.6 mg/kg | Dose Escalation: Cohort 3, 3.2 mg/kg | Dose Escalation: Cohort 4, 5.4 mg/kg | Dose Escalation: Cohort 5, 6.4 mg/kg | Dose Escalation: Cohort 6, 8.0 mg/kg | Dose Expansion: HER2-positive Breast Cancer, 5.4 mg/kg | Dose Expansion: HER2-positive Breast Cancer, 6.4 mg/kg | Dose Expansion: HER2-low Expressing Breast Cancer, 5.4 mg/kg | Dose Expansion: HER2-low Expressing Breast Cancer, 6.4 mg/kg | Dose Expansion: HER2-overexpressing Gastric or GEJ, 5.4 mg/kg | Dose Expansion: HER2-overexpressing Gastric or GEJ, 6.4 mg/kg | Dose Expansion: HER2-expressing Other Solid Tumors
Number analyzed (Participants) | 3 | 3 | 3 | 6 | 6 | 6 | 50 | 66 | 21 | 33 | 19 | 25 | 59
Participants
  Treatment-emergent adverse events (TEAEs) | 3 | 3 | 3 | 6 | 6 | 6 | 50 | 66 | 20 | 33 | 19 | 25 | 59
  Drug-related TEAEs | 3 | 2 | 2 | 6 | 6 | 6 | 50 | 66 | 20 | 33 | 18 | 25 | 59
  TEAEs ≥Grade 3 | 0 | 0 | 0 | 5 | 2 | 2 | 23 | 42 | 11 | 23 | 10 | 20 | 37
  Drug-related TEAEs ≥Grade 3 | 0 | 0 | 0 | 3 | 2 | 2 | 18 | 37 | 8 | 20 | 8 | 16 | 30
  Serious TEAEs (including AEs ending in death) | 0 | 0 | 0 | 1 | 1 | 1 | 11 | 17 | 3 | 12 | 4 | 7 | 18
  Drug-related serious TEAEs | 0 | 0 | 0 | 1 | 0 | 0 | 4 | 11 | 2 | 8 | 1 | 3 | 9
  TEAEs associated with death | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 1 | 0 | 2 | 0 | 1 | 5
  Drug-related TEAEs associated with death | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 2 | 0 | 0 | 2
  TEAEs associated with discontinuation of drug | 0 | 0 | 0 | 0 | 1 | 3 | 7 | 22 | 0 | 11 | 0 | 4 | 5
  Related TEAEs associated with drug discontinuation | 0 | 0 | 0 | 0 | 1 | 1 | 5 | 21 | 0 | 11 | 0 | 3 | 5
  TEAEs associated with dose reduction | 0 | 0 | 0 | 2 | 3 | 2 | 5 | 18 | 3 | 9 | 5 | 9 | 14
  Drug-related TEAEs associated with dose reduction | 0 | 0 | 0 | 2 | 3 | 2 | 4 | 18 | 2 | 9 | 4 | 9 | 13
  TEAEs associated with dose interruption | 1 | 1 | 0 | 6 | 4 | 3 | 21 | 36 | 8 | 13 | 9 | 13 | 22
  Related TEAEs associated with dose interruption | 1 | 0 | 0 | 3 | 3 | 2 | 15 | 28 | 7 | 11 | 5 | 11 | 17

ADVERSE EVENTS:
Time Frame: Treatment-emergent adverse event (TEAE) data were collected from baseline up to 28 days after the last dose of study drug, up to 3 years 5 months.
Description: TEAEs were AEs that occur, having been absent before the first dose of study drug, or has worsened in severity or seriousness after the first dose until 28 days after the last dose. Serious adverse events with an onset or worsening ≥29 days after the last dose, if related to the study treatment, are also TEAEs. TEAEs from other HER2-expressing solid tumors other than breast or gastric were combined as prespecified in the protocol (excluding 1 patient with gastric cancer who received 5.4 mg/kg).
Arm/Group | Dose Escalation: Cohort 1, 0.8 mg/kg | Dose Escalation: Cohort 2, 1.6 mg/kg | Dose Escalation: Cohort 3, 3.2 mg/kg | Dose Escalation: Cohort 4, 5.4 mg/kg | Dose Escalation: Cohort 5, 6.4 mg/kg | Dose Escalation: Cohort 6, 8.0 mg/kg | Dose Expansion: HER2-positive Breast Cancer, 5.4 mg/kg | Dose Expansion: HER2-positive Breast Cancer, 6.4 mg/kg | Dose Expansion: HER2-low Expressing Breast Cancer, 5.4 mg/kg | Dose Expansion: HER2-low Expressing Breast Cancer, 6.4 mg/kg | Dose Expansion: HER2-overexpressing Gastric or GEJ, 5.4 mg/kg | Dose Expansion: HER2-overexpressing Gastric or GEJ, 6.4 mg/kg | Dose Expansion: HER2-expressing Other Solid Tumors
All-Cause Mortality (participants affected / at risk) | 0/3 | 0/3 | 0/3 | 0/6 | 0/6 | 0/6 | 3/50 | 1/66 | 0/21 | 0/33 | 1/19 | 1/25 | 5/59
Serious Adverse Events (participants affected / at risk) | 0/3 | 0/3 | 0/3 | 1/6 | 1/6 | 1/6 | 11/50 | 17/66 | 3/21 | 12/33 | 4/19 | 7/25 | 18/59
Other Adverse Events (participants affected / at risk) | 3/3 | 3/3 | 3/3 | 6/6 | 6/6 | 6/6 | 50/50 | 66/66 | 20/21 | 33/33 | 19/19 | 25/25 | 59/59
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Dose Escalation: Cohort 1, 0.8 mg/kg (N=3) | Dose Escalation: Cohort 2, 1.6 mg/kg (N=3) | Dose Escalation: Cohort 3, 3.2 mg/kg (N=3) | Dose Escalation: Cohort 4, 5.4 mg/kg (N=6) | Dose Escalation: Cohort 5, 6.4 mg/kg (N=6) | Dose Escalation: Cohort 6, 8.0 mg/kg (N=6) | Dose Expansion: HER2-positive Breast Cancer, 5.4 mg/kg (N=50) | Dose Expansion: HER2-positive Breast Cancer, 6.4 mg/kg (N=66) | Dose Expansion: HER2-low Expressing Breast Cancer, 5.4 mg/kg (N=21) | Dose Expansion: HER2-low Expressing Breast Cancer, 6.4 mg/kg (N=33) | Dose Expansion: HER2-overexpressing Gastric or GEJ, 5.4 mg/kg (N=19) | Dose Expansion: HER2-overexpressing Gastric or GEJ, 6.4 mg/kg (N=25) | Dose Expansion: HER2-expressing Other Solid Tumors (N=59)
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 2 | 1 | 0
Cellulitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Sepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Lung infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Bacteraemia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Influenza (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Osteomyelitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Peritonitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Postoperative wound infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Pyelonephritis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Streptococcal bacteraemia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Soft tissue infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pneumocystis jirovecii pneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 0 | 0 | 3
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 3
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Contrast media allergy (Immune system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 1 | 0 | 3 | 2
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hypophosphataemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Tumour lysis syndrome (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Headache (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Peroneal nerve palsy (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Seizure (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Transient ischaemic attack (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Haematoma (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hypotension (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 2 | 0 | 3 | 0 | 1 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 0 | 0 | 1 | 0 | 0 | 1
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 0 | 0 | 0
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Colitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Diarrhoea haemorrhagic (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Dysphagia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Intestinal perforation (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Obstruction gastric (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pancreatitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Small intestine obstruction (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Stomatitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Mechanical ileus (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Gastrointestinal mucosa hyperaemia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Cholangitis (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1
Hepatic function abnormal (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Scleroderma-like reaction (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Cystitis haemorrhagic (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hydronephrosis (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Disease progression (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 1
Malaise (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Pyrexia (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Platelet count decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 0 | 2 | 0 | 1 | 2
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Blood alkaline phosphatase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Alanine aminotransferase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Blood bilirubin increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Troponin increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Humerus fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Radiation necrosis (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Central venous catheterisation (Surgical and medical procedures) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Dose Escalation: Cohort 1, 0.8 mg/kg (N=3) | Dose Escalation: Cohort 2, 1.6 mg/kg (N=3) | Dose Escalation: Cohort 3, 3.2 mg/kg (N=3) | Dose Escalation: Cohort 4, 5.4 mg/kg (N=6) | Dose Escalation: Cohort 5, 6.4 mg/kg (N=6) | Dose Escalation: Cohort 6, 8.0 mg/kg (N=6) | Dose Expansion: HER2-positive Breast Cancer, 5.4 mg/kg (N=50) | Dose Expansion: HER2-positive Breast Cancer, 6.4 mg/kg (N=66) | Dose Expansion: HER2-low Expressing Breast Cancer, 5.4 mg/kg (N=21) | Dose Expansion: HER2-low Expressing Breast Cancer, 6.4 mg/kg (N=33) | Dose Expansion: HER2-overexpressing Gastric or GEJ, 5.4 mg/kg (N=19) | Dose Expansion: HER2-overexpressing Gastric or GEJ, 6.4 mg/kg (N=25) | Dose Expansion: HER2-expressing Other Solid Tumors (N=59)
Nasopharyngitis (Infections and infestations) | 1 | 1 | 0 | 2 | 0 | 0 | 5 | 9 | 0 | 4 | 0 | 3 | 6
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 1 | 2 | 0 | 0 | 9 | 7 | 1 | 4 | 0 | 1 | 4
Cystitis (Infections and infestations) | 0 | 0 | 0 | 1 | 1 | 0 | 5 | 6 | 0 | 1 | 0 | 2 | 2
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 4 | 3 | 0 | 1 | 2 | 3 | 1
Influenza (Infections and infestations) | 0 | 1 | 0 | 2 | 0 | 1 | 3 | 3 | 1 | 0 | 1 | 1 | 2
Lung infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 3 | 0 | 1 | 1 | 2 | 1
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 2 | 0 | 2 | 0 | 0 | 3
Cellulitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 1 | 3 | 0 | 0 | 1
Conjunctivitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 3 | 1 | 0 | 1 | 1 | 0 | 1
Gastroenteritis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 1
Angular cheilitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 2 | 0
Bronchitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 1 | 0 | 0
Oral candidiasis (Infections and infestations) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 1
Anaemia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 3 | 2 | 1 | 23 | 30 | 7 | 14 | 4 | 14 | 23
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 1 | 3 | 0 | 1 | 3
Decreased appetite (Metabolism and nutrition disorders) | 2 | 1 | 1 | 4 | 4 | 2 | 23 | 47 | 7 | 20 | 8 | 22 | 35
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 9 | 13 | 1 | 6 | 4 | 3 | 9
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 5 | 9 | 2 | 6 | 0 | 4 | 5
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 9 | 1 | 2 | 0 | 3 | 5
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 3 | 0 | 0 | 0 | 0 | 7
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 2 | 2 | 0 | 1 | 0
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 2 | 0 | 0 | 2
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 2 | 0 | 0 | 2
Vitamin D deficiency (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0
Insomnia (Psychiatric disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 3 | 6 | 1 | 3 | 0 | 2 | 4
Anxiety (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 2 | 2 | 0 | 0 | 0 | 1
Dysgeusia (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 4 | 14 | 3 | 2 | 2 | 5 | 9
Headache (Nervous system disorders) | 2 | 0 | 0 | 0 | 0 | 0 | 8 | 11 | 0 | 4 | 4 | 0 | 4
Dizziness (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 8 | 5 | 3 | 4 | 0 | 1 | 8
Peripheral sensory neuropathy (Nervous system disorders) | 1 | 0 | 1 | 0 | 1 | 0 | 1 | 6 | 1 | 3 | 2 | 0 | 3
Neuropathy peripheral (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 3 | 2 | 0 | 1 | 0 | 1
Dry eye (Eye disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 6 | 8 | 2 | 1 | 1 | 0 | 1
Keratitis (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 5 | 0 | 1 | 0 | 0 | 1
Cataract (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 2 | 1 | 0 | 0 | 2 | 2
Vision blurred (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 3 | 0 | 2 | 0 | 0 | 1
Conjunctival haemorrhage (Eye disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 2 | 0 | 1 | 0 | 1 | 0 | 0
Retinal degeneration (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0
Retinal tear (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Macular fibrosis (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Tinnitus (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 1 | 0 | 1 | 0 | 0 | 1
Palpitations (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 2 | 0 | 2 | 0 | 0
Hypertension (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 2 | 0 | 4 | 0 | 1 | 0
Hypotension (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 5 | 0 | 1 | 0 | 0 | 1
Hot flush (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 2 | 0 | 2 | 0 | 0 | 0
Lymphoedema (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 0 | 0 | 1 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1 | 1 | 1 | 14 | 12 | 2 | 5 | 2 | 1 | 6
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 2 | 0 | 0 | 8 | 6 | 2 | 2 | 1 | 3 | 8
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 3 | 10 | 1 | 7 | 0 | 3 | 5
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 7 | 8 | 3 | 5 | 1 | 0 | 4
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 6 | 0 | 3 | 0 | 0 | 1
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 2 | 7
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 3 | 1 | 3 | 0 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 3 | 0 | 1 | 2 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 3 | 0 | 0 | 3
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 3 | 1 | 0 | 0 | 0 | 0
Organising pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 3 | 4 | 0 | 0 | 0 | 0 | 0
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 0 | 1 | 0 | 0 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 0 | 0 | 1 | 0 | 0 | 1
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 2 | 0 | 0 | 2
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 3 | 1 | 2 | 6 | 4 | 4 | 43 | 52 | 15 | 26 | 12 | 19 | 44
Vomiting (Gastrointestinal disorders) | 1 | 1 | 2 | 1 | 4 | 0 | 28 | 35 | 10 | 14 | 3 | 8 | 31
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 1 | 2 | 1 | 3 | 18 | 28 | 9 | 16 | 3 | 5 | 19
Constipation (Gastrointestinal disorders) | 0 | 0 | 1 | 4 | 2 | 1 | 18 | 30 | 7 | 14 | 5 | 7 | 16
Stomatitis (Gastrointestinal disorders) | 0 | 0 | 0 | 2 | 1 | 1 | 7 | 18 | 4 | 13 | 1 | 4 | 10
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 7 | 9 | 1 | 2 | 0 | 0 | 6
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 2 | 7 | 9 | 2 | 1 | 1 | 0 | 2
Abdominal distension (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 3 | 0 | 3 | 8 | 1 | 1 | 0 | 0 | 1
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 5 | 1 | 2 | 0 | 0 | 2
Flatulence (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 3 | 3 | 1 | 0 | 0 | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 3 | 1 | 1 | 1 | 0 | 0 | 2
Ascites (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 2 | 1 | 0 | 0 | 1 | 3
Dry mouth (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 4 | 1 | 0 | 0 | 0 | 1
Abdominal discomfort (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 1 | 0 | 1 | 0 | 0 | 0
Gingival bleeding (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 3 | 0 | 1 | 2 | 0 | 0 | 0
Haemorrhoids (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 0 | 3 | 0 | 0 | 0
Gastritis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 2 | 0 | 0 | 1
Toothache (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 1 | 1 | 0 | 1
Faeces discoloured (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0
Periodontal disease (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Hepatic function abnormal (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 3 | 2
Cholangitis (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 2 | 3 | 3 | 19 | 45 | 6 | 18 | 4 | 4 | 20
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 5 | 8 | 1 | 4 | 1 | 1 | 6
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 6 | 8 | 0 | 5 | 1 | 0 | 2
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 6 | 1 | 1 | 0 | 1 | 3
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 4 | 4 | 0 | 1 | 2 | 1 | 2
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 2 | 1 | 1 | 0 | 0 | 0 | 4
Nail disorder (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 4 | 0 | 2 | 1 | 0 | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 3 | 1 | 0 | 2 | 0 | 1 | 0
Erythema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 1 | 0 | 0
Onychoclasis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0
Rash erythematous (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Madarosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 5 | 6 | 2 | 2 | 0 | 2 | 4
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 3 | 6 | 1 | 2 | 1 | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 4 | 1 | 4 | 0 | 0 | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 2 | 1 | 1 | 1 | 0 | 2
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 2 | 1 | 0 | 0 | 0 | 3
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 5 | 1 | 0 | 0 | 0 | 1
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 2 | 0 | 0 | 0 | 0 | 0
Fatigue (General disorders) | 3 | 0 | 0 | 0 | 3 | 4 | 24 | 32 | 11 | 9 | 4 | 3 | 21
Malaise (General disorders) | 0 | 0 | 0 | 2 | 0 | 1 | 6 | 19 | 2 | 13 | 3 | 5 | 13
Pyrexia (General disorders) | 1 | 0 | 1 | 2 | 0 | 0 | 10 | 18 | 1 | 9 | 3 | 8 | 9
Oedema peripheral (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 10 | 10 | 4 | 4 | 2 | 1 | 6
Oedema (General disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 3 | 7 | 0 | 1 | 1 | 4 | 2
Chills (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 6 | 5 | 0 | 1 | 0 | 0 | 0
Influenza-like illness (General disorders) | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 5 | 0 | 1 | 0 | 0 | 1
Pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 2 | 0 | 1 | 0 | 0 | 1
Asthenia (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 1 | 0 | 0 | 0 | 0 | 0
Chest discomfort (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0
Platelet count decreased (Investigations) | 0 | 0 | 1 | 4 | 3 | 3 | 15 | 24 | 3 | 14 | 5 | 12 | 22
Neutrophil count decreased (Investigations) | 0 | 1 | 0 | 4 | 2 | 1 | 12 | 25 | 3 | 13 | 2 | 12 | 21
White blood cell count decreased (Investigations) | 0 | 1 | 0 | 3 | 2 | 1 | 9 | 22 | 4 | 13 | 3 | 11 | 17
Aspartate aminotransferase increased (Investigations) | 0 | 1 | 1 | 2 | 1 | 0 | 9 | 23 | 3 | 10 | 1 | 3 | 12
Alanine aminotransferase increased (Investigations) | 0 | 0 | 0 | 1 | 1 | 0 | 7 | 17 | 1 | 7 | 1 | 3 | 8
Weight decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 5 | 9 | 3 | 5 | 2 | 0 | 11
Blood alkaline phosphatase increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 5 | 7 | 0 | 4 | 2 | 1 | 7
Electrocardiogram QT prolonged (Investigations) | 2 | 0 | 0 | 1 | 0 | 0 | 5 | 6 | 4 | 1 | 1 | 0 | 1
Lymphocyte count decreased (Investigations) | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 8 | 0 | 2 | 0 | 4 | 2
Blood creatinine increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 3 | 1 | 4 | 4
Blood bilirubin increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 7 | 0 | 2 | 1 | 1 | 0
Weight increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 3 | 6 | 0 | 1 | 0 | 0 | 1
Blood lactate dehydrogenase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 3 | 1 | 1 | 1 | 0 | 0 | 0
Ejection fraction decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 5
Protein total decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 2 | 0 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 3 | 1 | 2 | 1 | 0 | 1
Infusion-related reaction (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 2 | 1 | 0 | 1 | 0 | 0
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Herpes zoster (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 2 | 0 | 1 | 0 | 1 | 1
Paronychia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 2 | 0 | 1 | 0 | 0 | 2
Pharyngitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 2 | 0 | 1 | 0 | 1 | 1
Sinusitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 1
Ear infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Oral herpes (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Folliculitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Soft tissue infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Mucosal infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 2 | 1 | 1 | 0 | 0 | 0
Tumour-associated fever (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Haemangioma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cold type haemolytic anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Depression (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 0 | 0 | 0 | 0 | 0
Retinal haemorrhage (Eye disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 0 | 2
Corneal disorder (Eye disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 1
Vitreous floaters (Eye disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Uveitis (Eye disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vertigo (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 1
Tachycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 3 | 1 | 1 | 0 | 0 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 3 | 0 | 2 | 0 | 0 | 3
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Eructation (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Dental caries (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Intestinal perforation (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 2 | 0 | 0 | 0 | 0 | 2
Nail discolouration (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 2 | 0 | 0 | 0 | 0 | 0
Haemorrhage subcutaneous (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Xeroderma (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 2 | 2 | 0 | 1 | 0 | 0 | 1
Joint stiffness (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Osteoporosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Blood creatinine phosphokinase increased (Investigations) | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Thermal burn (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-04-26): https://cdn.clinicaltrials.gov/large-docs/00/NCT02564900/Prot_SAP_000.pdf